CLINICAL TRIAL: NCT05894356
Title: The Paternal Clock: Uncovering the Consequences of Advanced Paternal Age on Sperm DNA Fragmentation
Acronym: Paternal Clock
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3287
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men undergoing sperm DNA fragmentation test: Men presenting at the clinic for infertility evaluation
  Interventions: Other: Study chart review

INTERVENTIONS:
Other: Study chart review — Evaluation of 4250 sperm DNA fragmentation samples with the goal of defining a cut-off age beyond which SDF levels increase significantly

SUMMARY:
Sperm DNA fragmentation (SDF) serves as a marker for chromatin and DNA damage in sperm. Assessing sperm DNA integrity is crucial in male fertility evaluation since high levels of SDF are associated with a greater number of adverse reproductive outcomes, including an increased risk of miscarriage and birth defects.

Recent research suggests that advanced paternal age (APA) may lead to DNA damage in sperm, however the precise age at which this risk becomes apparent has not yet been clearly defined, necessitating the identification of the point in time at which high SDF levels occur. With the help of this knowledge, male infertility can be diagnosed with greater accuracy, and infertile couples can receive appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Male of at least 18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sperm sample
Study Population: Male patients presenting for infertility evaluation from all ages, ethnicities, and medical histories.
Sampling Method: Non-Probability Sample
Enrollment: 4250 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Investigate the impact of advanced paternal age on sperm DNA fragmentation | Up to 3 weeks
  Comparing mean sperm DNA fragmentation throughout the chart review of different age groups

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No